CLINICAL TRIAL: NCT04390464
Title: mulTi-Arm Therapeutic Study in Pre-ICu Patients Admitted With Covid-19 - Repurposed Drugs (TACTIC-R)
Acronym: TACTIC-R
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Frances Hall, Consultant Rheumatologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACTIC-R
Record Dates: First submitted 2020-05-08; First posted 2020-05-15 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — ravulizumab; baricitinib; Standard of Care

STUDY DESIGN:
Intervention Model Description: TACTIC-R is a randomised, parallel arm, open-label platform trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (Active Comparator): Standard of care
  Interventions: Other: Standard of care
- Ravulizumab + Standard of care (Experimental): Ravulizumab IV (adjusted to weight, Day 1 only)
  Interventions: Drug: Ravulizumab
- Baricitinib + Standard of care (Experimental): Baricitinib PO OD (4mg, Days 1-14)
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Ravulizumab — Ravulizumab (Ultomiris, Alexion Pharmaceuticals) is a monoclonal antibody that binds to terminal complement protein C5 and prevents the complement-mediated destruction of cells. It is administered by intravenous infusion. Ravulizumab has a marketing authorisation in the UK for treating Paroxysmal Nocturnal Haemoglobinuria in adults.
  Other Names: Ultomiris
  Arms: Ravulizumab + Standard of care
Drug: Baricitinib — Baricitinib is administered orally once daily. It is licensed for treatment of rheumatoid arthritis, it is a relatively fast acting disease modifying anti-rheumatic drug and has the potential to be scaled up for use for a pandemic.
  Other Names: Olumiant
  Arms: Baricitinib + Standard of care
Other: Standard of care — Regular standard of care for COVID-19 patients
  Arms: Standard of care

SUMMARY:
TACTIC-R is a randomised, parallel arm, open-label platform trial for investigating potential treatment for COVID-19 disease. While SARS-CoV infection evades detection by the immune system in the first 24 hours of infection, it ultimately produces a massive immune system response in the subgroup of people who develop severe complications. Most tissue damage following infection with COVID19 appears to be due to a later, exaggerated, host immune response. This leads to lung and sometimes multi-organ damage.

Most people who develop these severe complications still have virus present in their respiratory tract at the time-point when the disease starts to evolve. Immune modulation in the presence of active infection has potential to cause more harm than benefit. Safety considerations when studying immune modulation strategies are paramount. Therefore, this study proposes to assess the efficacy of immunomodulatory agents that target dysregulated immune response that drive the severe lung, and other organ, damage. The medications investigated for efficacy in this trial are Baricitinib and Ravulizumab.

DETAILED DESCRIPTION:
TACTIC-R will assess the efficacy of the immunomodulatory agents Baricitinib and Ravulizumab as potential treatments for COVID-19 disease against Standard of Care alone. These agents target the dysregulated immune response that drives the severe lung, and other organ, damage frequently seen during COVID-19 infection. This trial will compare these immunomodulatory agents to Standard of Care over a 14-day treatment period, with follow-up at 28 and 90 days. Patients will be randomised in a 1:1:1 ratio across treatments.

TACTIC-R will use a platform design with interim analysis to make efficient decisions about efficacy and futility (e.g. lack of efficacy and risk of harm) of the trial treatments. This enables the trial to stop recruiting to arms early where a clear efficacy decision can be made. It also allows for the addition of further arms.

TACTIC-R will also iterate an algorithm for use of clinical and biochemical phenotyping to:

1. Stratify patients to therapeutic arms according to probability of efficacy
2. Identify early indicators of failure of therapeutic strategy.

By collecting samples for genomics, transcriptomics, proteomics and immunological phenotyping, parallel studies associated with TACTIC-R will investigate host susceptibility factors for development of severe COVID-19-related disease and predictive biomarkers of response to therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria

To be included in the trial the participant must:

1. Be aged 18 and over
2. Have clinical picture strongly suggestive of COVID-19-related (with/without positive COVID-19 test) AND

   * Risk count (as defined below) >3 OR
   * ≥ 3 if risk count includes "Radiographic severity score >3"
3. Be considered an appropriate subject for intervention with immunomodulatory in the opinion of the supervising clinician
4. Be able to be maintained on venous thromboembolism prophylaxis or current maintenance therapy during inpatient dosing period, according to local guidelines

Exclusion Criteria

The presence of any of the following will preclude participant inclusion:

1. Inability to supply direct informed consent or assent from Next of Kin or Independent Healthcare Provider on behalf of patient
2. Mechanical ventilation at time of prior to dosing
3. Contraindications to study drugs, including hypersensitivity to the active substances or any of the excipients
4. Currently on any of the study investigational medicinal products
5. Known unresolved Neisseria meningitidis infection
6. Unwilling to be vaccinated against Neisseria meningitidis or receive prophylactic antibiotic cover until 2 weeks after vaccination
7. Known active tuberculosis (no blood screening required)
8. Known active Hepatitis B or C (no blood screening required); active varicella zoster
9. Concurrent participation in any interventional clinical trial including COVID-19-related disease trials (observational studies allowed)
10. Patient moribund at presentation or screening
11. Pregnancy at screening (or unwillingness to adhere to pregnancy advice in protocol)
12. Unwillingness to adhere to breastfeeding advice in protocol
13. Either alanine transaminase or aspartate transaminase (ALT or AST) > 5 times the upper limit of normal
14. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. Cockcroft Gault estimated creatinine clearance < 30 ml /min/1.73 m^2)
15. Currently receiving probenecid or chronic IVIG treatment
16. Any medical history or clinically relevant abnormality that is deemed by the principal investigator and/or medical monitor to make the patient ineligible for inclusion because of a safety concern.

Risk Count

Patients will be given a Risk Count equal to the cumulative points received for the following criteria (no = 0 points, yes = 1 point):

Male gender, Age > 40 years, Non-white ethnicity, Diabetes, Hypertension, Neutrophils > 8.0x10^9/L, CRP > 40mg/L, Radiographic severity score >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1167 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-05-07 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to incidence of the composite endpoint of: Death, Mechanical ventilation, ECMO, Cardiovascular organ support, or Renal failure | up to Day 14
  Number of days taken for occurrence of one of the following events: 1. Death 2. Mechanical ventilation 3. Extracorporeal membrane oxygenation (ECMO) 4. Cardiovascular organ support (balloon pump or inotropes) 5. Renal failure (estimated creatinine clearance (by Cockcroft-Gault formula) <15 ml /min/1.73m^2), haemofiltration or dialysis

SECONDARY OUTCOMES:
Change in clinical status as assessed on 7-point ordinal scale compared to baseline | 14 days
  The clinical status of the patients is assessed using 7-point ordinal scale as follows: 1 = Death, 2 = Mechanical ventilation, 3 = Non-invasive or high flow oxygen, 4 = Low flow oxygen, 5 = Hospitalised - no oxygen, 6 = Discharged - normal activities not resumed, 7 = Discharged - normal activities resumed
Proportion of patients with adverse events of special interest in each treatment arm | 14 days
  The proportion of patients in each treatment arm that experience adverse events of special interest, defined as: venous thromboembolism, new infections requiring antimicrobials
Time to Sp02 >94% on room air | 14 days
  The time taken to achieve blood oxygen saturation levels above 94% in patients on room air, measured in hours/days
Time to first negative SARS-CoV2 PCR | 14 days
  The amount of time between a patient's first positive SARS-CoV2 PCR test and a patient's first negative SARS-CoV2 PCR test, measured in days
Duration of oxygen therapy | 14 days
  The duration of oxygen therapy given to a patient, measured in days
Duration of hospitalisation | 14 days
  The duration of hospitalisation of a patient, measured in days
All cause mortality at day 28 | 28 Days
  The number of deaths recorded at 28 days irrespective of the cause
Time to clinical improvement | 14 days
  The time to clinical improvement for a patient, defined as: >2 point improvement from Day 1 on the 7-point ordinal scale, measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Frances Hall Hall, FRCP (UK), D.Phil, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Hall FC, Cheriyan J, Cope AP, Galloway J, Wilkinson I, Bond S, Norton S, Banham-Hall E, Bayes H, Kostapanos M, Nodale M, Petchey WG, Sheeran T, Underwood J, Jayne DR; TACTIC-R Investigators Group. Efficacy and safety of baricitinib or ravulizumab in adult patients with severe COVID-19 (TACTIC-R): a randomised, parallel-arm, open-label, phase 4 trial. Lancet Respir Med. 2023 Dec;11(12):1064-1074. doi: 10.1016/S2213-2600(23)00376-4. Epub 2023 Nov 14. PMID 37977159
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Kulkarni S, Fisk M, Kostapanos M, Banham-Hall E, Bond S, Hernan-Sancho E, Norton S, Cheriyan J, Cope A, Galloway J, Hall F, Jayne D, Wilkinson IB. Repurposed immunomodulatory drugs for Covid-19 in pre-ICu patients - mulTi-Arm Therapeutic study in pre-ICu patients admitted with Covid-19 - Repurposed Drugs (TACTIC-R): A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jul 8;21(1):626. doi: 10.1186/s13063-020-04535-4. PMID 32641154